CLINICAL TRIAL: NCT05300360
Title: Prospective Observational Study Evaluating the Prevalence of Adenosine Deaminase (ADA) Enzyme Deficiency Disease in Adult Patients With Pulmonary Alveolar Proteinosis in Pulmonology Clinics
Brief Title: Prevalence of Adenosine Deaminase (ADA) Enzyme Deficiency Disease in Adult Patients With Pulmonary Alveolar Proteinosis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: TRPHARM (Industry)
Responsible Party: Sponsor
Other Study IDs: TR-ADA-006
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Alveolar Proteinosis
Keywords: Pulmonary Alveolar Proteinosis, adenosine deaminase, guithre paper
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: adenosine deaminase test — adenosine deaminase enzyme deficiency test

SUMMARY:
This observational study was designed as a prospective epidemiological screening study. Patients who have applied to the centers participating in the study and who have previously been clinically or pathologically diagnosed with PAP (Pulmonary alveolar proteinosis) will be included in the study. Up-to-date data will be collected from patients who have agreed to participate in the study, and a blood sample with DBS will be taken from patients. The blood taken will be subjected to analysis for ADA metabolites. For patients with a high metabolic test, the responsible researcher will advise on clarifying the diagnosis with a genetic test other than the study. In case of formation of new information for each patient, consultation will be provided by the responsible researcher. Thus, the prevalence of ADA enzyme deficiency disease will be evaluated in patients diagnosed with PAP.

DETAILED DESCRIPTION:
PAP (Pulmonary alveolar proteinosis) is a rare disease with a frequency of 0.36 per million. As a result of intensive accumulation of surfactant components in the lungs, it leads to respiratory distress at various levels. PAP has been frequently monitored among patients with ADA enzyme deciency. Primary immunodeficiency diseases are a group of diseases that are accompanied by chronic and/or recurrent bacterial, fungal, protozoal and viral infections that develop as a result of primary or congenital immunodeficiency. The incidence dec in society varies from 1/10,000 to 1/100,000. Combined immunodeficiencies account for 15-29% of primary immunodeficiencies. Severe Combined Immunodeficiencies (SCID) are a heterogeneous group of diseases caused by hereditary errors in genes involved in the development and/or function of T, B, and sometimes NK cells, which cause serious dysfunction of the immune system. The incidence is estimated at 1/100,000 live births in the United States. Although the exact incidence of inbreeding is not known in our country, where inbreeding is common, it is expected that those who show autosomal recessive transition will be more common, especially. The recognition of these disorders by clinicians is important for reducing long-term complications due to recurrent infections and preventing mortality with appropriate treatment. The frequency of SCIDY in our country is unknown. Unlike in Europe and America, SCID types, which are autosomal recessive in our country, are considered to be the most common form due to the high rates of inbreeding. The ratio obtained by comparing the number of live babies born in a year in Konya with the number of SCID cases diagnosed in the same year in the Pediatric Immunology Clinic of the Meram Faculty of Medicine of Selcuk University, the only primary immunodeficiency diagnostic center in the region, is 1/10,000. This preliminary study shows that in our country this disease is much more common than in Europe and America. To date, more than 20 genetic defects have been identified that cause SCID. All known genetic defects disrupt the development of cells of the immune system, causing combined immunodeficiency. One of them, the ADA defect, is also a metabolic disease, due to which there is a lack of enzymes. ADA catalyzes the deamination of purine nucleosides adenosine (Ado) and 2'-deoxyadenosine (dAdo), which are produced during the degradation and transformation of RNA and DNA. ADA is a cleansing enzyme: it detoxifies purines. In ADA deficiency, 2'-deoxyadenosine (dAdo) is phosphorylated and converted into deoxyadenosine triphosphate (dATP). Accumulation of DATP disrupts DNA repair and replication. In ADA deficiency, a high percentage of dATP accumulates, especially in erythrocytes and lymphocytes. Increased levels of adenosine break down the wall of the lymphocyte. It inhibits the development of lymphocytes in the thymus. A kind of lymphocyte intoxication occurs. It leads to a severe form of lymphopenia. Approximately 10-20% of SCID are diagnosed as ADA enzyme deficiency. It shows an autosomal recessive transition. Your gene is 20. it is localized on the long arm of the chromosome.

Clinically, there are early and late onset types:

Classic-early onset ADA deficiency: Although normal at birth, patients present with infections seen from the first months of life, resulting in death if left untreated. In addition to the AKI table, neuro-developmental disorders, sensorineural hearing loss and/or skeletal abnormalities have also been reported in these patients. Although hematopoietic stem cell transplantation, enzyme replacement therapy and gene therapy are treatment approaches that provide cure, early diagnosis determines the prognosis.

Late-onset ADA deficiency: Patients may present with recurrent infections, bronchiectasis, autoimmunity, human papillomavirus (HPV) infections at an older age, even in adulthood. Lymphopenia is an invariable finding. High IgE and eosinophilia may be observed. In these cases, residual enzyme activity due to the type of mutation causes a late onset. This phenotype accounts for 10-15% of all cases of ADA deficiency.

Patients with late-onset ADA enzyme deficiency appear in the form of case reports. in a study in which the data of two patients were shared in Zurich in 1997, one patient had a history of recurrent otitis and pulmonary infection, bronchiectasis, lymphopenia, and immunoglobulin E elevation. The other patient, his cousin ADA, was diagnosed by chance while undergoing a bone marrow scan due to enzyme deficiency. He had a history of recurrent tonsillitis.

In a study conducted by Hacettepe University published in 2018. The data of 13 ADA enzyme deficient patients were evaluated and it was determined that 3 patients with late/delayed diagnosis had ADA enzyme deficiency. A patient with a late diagnosis of ADA enzyme deficiency was found to have recurrent pneumonia, bronchiectasis, and immunoglobulin E elevation.

In the study in which the data of a patient with a late onset ADA enzyme deficiency published in Konya from our country in 2010 were shared, it was observed that the patient had a history of resection of the lower left lobe due to bronchiectasis, lymphopenia and an increase in immunoglobulin E.

Diagnosis: ADA enzyme deficiency is included in severe combined immunodeficiencies and is observed with lymphopenia and infections. The diagnosis is made by measuring the activity of the enzyme ADA in erythrocytes or lymphocytes in patients with suspected clinical and laboratory features (such as lymphopenia, bronchiectasis). By mutation analysis, a gene defect is shown. However, T-cell receptor excision circles (TREC) test is used for early diagnosis. However, since the TREC test is found to be normal at birth in late-onset patients, screening that leads patients to an early diagnosis can only be achieved by measuring ADA metabolites.

In late-onset ADA deficiency, it is difficult to diagnose. Low awareness of the disease and its symptoms usually results in these cases not being diagnosed, not being able to reach effective treatment, permanent organ damage and patient loss. For this reason, diagnosis of patients is very important in terms of quality of life, as well as vital importance.

Reason ADA enzyme deficiencies account for approximately 15% of severe combined immunodeficiencies. In 15-20% of patients with ADA enzyme deficiency, ADA enzyme deficiency is observed with a late diagnosis. Because of the inability of these patients to get a diagnosis, their treatment is also inadequate. For the first time in our country, this study aims to determine the diagnosis and obtain preliminary data on the prevalence of ADA disease by looking at ADA metabolites in a group of adult patients diagnosed with PAP.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the written informed consent form by the patient and/or his legal representative,
2. The patient should be between the ages of 18 and 70,
3. Diagnosis of PAP: The patient has been diagnosed with PAP clinically or histologically.

Exclusion Criteria:

* The patient was diagnosed with ADA enzyme deficiency before being included in the study,
* The patient's PAP diagnosis is secondary to an occupational disease such as silicosis,
* The patient's PAP diagnosis is secondary to an oncological disease,
* The patient has participated in an interventional clinical trial within the last 30 days,
* The patient himself and/or his legal representative did not give their consent to participate in the study,
* According to the researcher's opinion, the patient will not be able to properly fulfill the study requirements,

  * Pregnancy and/or lactation period,
* The fact that the volunteer participating in the study received an erythrocyte suspension or a complete blood transfusion within the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: male and female patients aged 18-70
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2022-08-16 (Estimated)

PRIMARY OUTCOMES:
The rate of ADA enzyme deficiency in PAP patients | six months
  The proportion of adult patients with PAP who are above the ADA metabolite test threshold and are suspected of having ADA enzyme deficiency.

SECONDARY OUTCOMES:
e ratio of PAP and ADA enzyme deficiency | 6 months
  The relationship between the level and frequency of lymphopenia and ADA enzyme dec disease
The relationship between lymphopenia and ADA enzyme deficiency | 6 months
  The relationship between the level and frequency of lymphopenia and ADA enzyme deciency disease
graphic parameters with lymphopenia | 6 months
  The relationship between lymphopenia and demograpfic parameters
Family history and ADA | 6 months
  Family history of immunodeficiency/ADA
The presence of inbreeding and the relationship of adenosine deaminase | 6 months
  The presence of inbreeding
The rate of late ADA enzyme deficiency disease | 6 months
  The rate of late ADA enzyme deficiency disease
infection frequency and ADA enzyme deficiency | 6 months
  The relationship between infection frequency and ADA enzyme deficiency

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Yedikule Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Maltepe, Turkey (Türkiye)